CLINICAL TRIAL: NCT07051915
Title: Comprehensive Evaluation of Two Second-Line Therapeutic Approaches for Immune Thrombocytopenia (ITP) - a Pragmatic Randomized Controlled Trial
Brief Title: The Holistic Study
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: Oslo University Hospital (Other); University Hospital, Akershus (Other); Sykehuset i Vestfold HF (Other); St. Olavs Hospital (Other); Helse Stavanger HF (Other Government); Sorlandet Hospital HF (Other Government); University Hospital of North Norway (Other); Haukeland University Hospital (Other); Helse Nord-Trøndelag HF (Other); Helse Fonna (Other); Nordlandssykehuset HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RGCH006
Record Dates: First submitted 2025-06-23; First posted 2025-07-04 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Thrombocytopenia Purpura
Keywords: Avatrombopag; Rituximab; Thrombocytopenia; Immune thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic; Thrombocytopenia; Purpura, Thrombocytopenic, Idiopathic | interventions — avatrombopag; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Avatrombopag (Experimental): Open label, oral Avatrombopag 20 mg tablets taken daily during the first week. Dose tapering period commencing from week 28 for up to 8 weeks.
  Interventions: Drug: Avatrombopag; Drug: Rituximab (Arm B)
- Rituximab (Active Comparator): Open label, intravenous infusions of 1000mg Rituximab 2 weeks apart
  Interventions: Drug: Avatrombopag; Drug: Rituximab (Arm B)

INTERVENTIONS:
Drug: Avatrombopag — Daily tablets
Drug: Rituximab (Arm B) — I.V.

SUMMARY:
This study is a phase 3 study where eligible patients will be randomized 1:1 to one of two treatment strategies: receiving a thrombopoietin receptor agonist (Avatrombopag), or anti-CD20 (Rituximab).

DETAILED DESCRIPTION:
This is a multi-center, international, open label randomized, controlled pragmatic trial consisting of 3 phases:

1. First phase extends from randomization to week 28
2. Second phase extends from week 28 to 78
3. Third phase extends from week 78 to the end of the trial (i.e. the last patient completing week 78)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 years.
2. Diagnosis of primary ITP of less than one-year duration and having a platelet count of < 30 x109/L measured within two weeks prior to inclusion with failure to achieve response or relapse after at least one cycle of dexamethasone (20-40 mg daily for 4 days) or prednisone /prednisolone (1 mg/kg for at least two weeks). Shorter courses or lower doses are allowed if discontinued or modified due to side effects.
3. Clinical need for subsequent platelet elevating therapy assessed by the physician in charge.
4. Signed and dated written informed consent.

Exclusion Criteria:

1. Previous treatment for ITP with: Rituximab, other immune suppressants (including mycophenolate mofetil, azathioprine, cyclosporine), dapsone, danazol, chemotherapy (apart from vincristine as rescue therapy) or splenectomy. Short treatment with any thrombopoietic agent is allowed if given for a limited duration of a maximum of 2 weeks as rescue therapy for quick elevation of platelet count in emergency situations e.g. bleeding.
2. Pregnancy or lactation.
3. Females of child-bearing potential refusing to follow effective contraceptive methods for at least 12 months following the last administration of Rituximab or during treatment with Avatrombopag.
4. Secondary ITP: ITP secondary to lymphoma or chronic lymphocytic leukemia; ITP secondary to the following autoimmune disorders: Systemic Lupus Erythematosus, Antiphospholipid Syndrome, or Common Variable Immune Deficiency; ITP secondary the following viral infections: Human Immunodeficiency Virus or Hepatitis C Virus.
5. Concomitant autoimmune hemolytic anemia.
6. Active hepatitis B virus (positive HBsAg). Patients with HBsAg negative and HBV core antigen antibody positive (HBcAb) should accept to receive entecavir (Baraclude) for 12 months if they will be allocated to Rituximab. Monthly HBV DNA monitoring will be required while on treatment and for the 6 months after the last dose of the study drug.
7. Presence of any serious comorbidity where the condition may worsen by and of the study drugs.
8. Known allergy, sensitivity or contraindication to Rituximab or Avatrombopag.
9. Patients in a severely immune compromised state.
10. Presence of active malignancy unless deemed cured by adequate treatment. Participants with the following neoplastic conditions can be included:

    1. Monoclonal gammopathy of undetermined significance (MGUS) or monoclonal B lymphocytosis of undetermined significance (MBUS).
    2. Basal/squamous cell carcinoma of the skin
    3. Carcinoma in situ of the cervix
    4. Carcinoma in situ of the breast
    5. Incidental histological finding of prostate cancer (TNM stage T1a or T1b).
11. Patients with history of poor compliance or history of alcohol/drug abuse or excessive alcohol beverage consumption that would interfere with the ability to comply with the study protocol, or current or past psychiatric disease that might interfere with the ability to comply with the study protocol or give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the oral TPO-RA, Avatrombopag, to Rituximab | Assessed at week 28
  To compare the efficacy of the oral TPO-RA, Avatrombopag to Rituximab by measuring the rates of durable responses defined as achieving platelet counts ≥ 50 X109/L in ≥3 of the bi-weekly measurements between weeks 20 and 28 including the last count without having received any other platelet elevating agents after randomization apart from rescue therapy received before end of week 10.

SECONDARY OUTCOMES:
The changes in the disease specific HRQoL | Baseline to weeks 28 and weeks 78
  The changes in the disease specific HRQoL from baseline to weeks 28 and 78 measured by ITP-PAQ (Overall Quality of Life Scale) score.
Changes in the level of fatigue | Baseline to weeks 28 and weeks 78
  The changes in the level of fatigue from baseline to weeks 28 and 78 measured by FACIT-Fatigue score
Rates of Sustained Response Off-Treatment (SROT) | At 78 weeks
  The rates of Sustained Response Off-Treatment (SROT) at 78 weeks where the occurrence of SROT defined as
  * A platelet count > 50 X109/L in at least 3 of the 4 planned visits between weeks 36 and 78 including week 78
  * No administration of platelet elevating agent between weeks 36 and 78.